CLINICAL TRIAL: NCT03371602
Title: Study of the Combined Influence of Sepsis and Mechanical Ventilation on the Human Diaphragm
Acronym: SEPTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL15_0423
Record Dates: First submitted 2017-10-03; First posted 2017-12-13 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Experimental): non-septic mesocolic programmed abdominal or thoracic surgery: gastrectomy, esophagectomy, pancreatectomy, hepatectomy
  Interventions: Procedure: surgery
- sepsis group (Experimental): Abdominal or thoracic surgery in a septic context (peritonitis, mediastinitis, pleural abscess)
  Interventions: Procedure: surgery
- mechanical ventilation group (Experimental): Patient in brain death for whom a multi-organ sampling is planned
  Interventions: Procedure: multi-organ sampling
- mechanical ventilation - sepsis group (Experimental): Patient under controlled mechanical ventilation to undergo abdominal or thoracic surgery in a septic context (peritonitis, mediastinitis, pleural abscess)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — a diaphragmatic biopsy (100 microgram) and a parietal biopsy will be performed by the surgeon during surgery.
  Arms: control group; mechanical ventilation - sepsis group; sepsis group
Procedure: multi-organ sampling — a diaphragmatic biopsy (100 microgram) will be performed by the surgeon during surgery.
  Arms: mechanical ventilation group

SUMMARY:
The aim of this study is to study the combined impact of mechanical ventilation and sepsis on the human diaphragm in order to establish the neutral, protective or destructive character of mechanical ventilation by studying the diameter of the fibers, activation of proteolytic systems, inhibition of protein synthesis, tissue inflammation as well as contractile function.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age, male or female requiring abdominal or thoracic surgery or multi-organ sampling;
* Affiliated to a social security or similar system;
* Not subject to legal protection;
* Having given consent to participate in the study (or consent from the trusted person)
* Control group (C): non-septic mesocolic programmed abdominal or thoracic surgery: gastrectomy, esophagectomy, pancreatectomy, hepatectomy
* Sepsis group (S): Abdominal or thoracic surgery in a septic context (peritonitis, mediastinitis, pleural abscess)
* Group Mechanical Ventilation (MV): Patient in brain death for which a multi organ sample is planned
* Mechanical Ventilation + Sepsis (S-MV) group: Patient under controlled mechanical ventilation to undergo abdominal or thoracic surgery in a septic context (peritonitis, mediastinitis, pleural abscess)

Exclusion Criteria:

* Pregnant woman (diagnosis of interrogation)
* severe and / or unbalanced chronic respiratory disease; severe malnutrition
* Long-term corticosteroids> 5mg / day for more than 1 month
* Myopathy
* surgery by laparoscopic

By group:

* Control group: Sepsis, preoperative controlled mechanical ventilation and preoperative hemodynamic instability
* Mechanical Ventilation Group: Sepsis, duration of controlled mechanical ventilation <24 hours or> 7 days
* Sepsis Group: Preoperatively controlled mechanical ventilation
* Mechanical Ventilation - Sepsis Group: duration of controlled mechanical ventilation <24 hours or> 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Assessment of atrophy of the myofibers of the human diaphragm | day 0 (day of the surgery)
  Atrophy of the myofibers will be assessed by comparison of the cross sectional area of the three different types of myofibers between the sepsis-mechanical ventilation group and the sepsis group, the ventilation group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Céline Guichon, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix Rousse Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: No